CLINICAL TRIAL: NCT02493036
Title: A Single-Dose, Open-Label, Extension Study to Evaluate the Sustainability of the Effects of SYN-010 in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: A Single-Dose, Open-Label, Study to Evaluate the Sustainability of the Effects of SYN-010 in Patients With IBS-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-2-010-002
Record Dates: First submitted 2015-06-29; First posted 2015-07-09 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)

STUDY DESIGN:
Intervention Model Description: Subjects from the study SB-2-010-001 (NCT02495623) were given either SYN-010 21 mg, SYN-010 42 mg, or Placebo. The subjects were offered the opportunity to roll over into SB-2-010-002 and receive SYN-010 42 mg. Some of the analyses were done from day one of SYN-010-001.
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Dose SYN-010 (Experimental): 42-mg SYN-010
  Interventions: Drug: SYN-010

INTERVENTIONS:
Drug: SYN-010

SUMMARY:
A Single-Dose, Open-Label, Extension Study to Evaluate the Sustainability of the Effects of SYN-010 in Patients with Irritable Bowel Syndrome with Constipation

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, open-label study. Up to sixty subjects with irritable bowel syndrome with constipation who are between the ages of 18 and 65, inclusive, will be enrolled. Subjects must have completed the previous SB-2-010-001 study. The entire duration of the study may be up to 57 days (from enrollment to the post end-of-study [EOS] visit telephone call).

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed Study SB-2-010-001.
* Subject must be willing to abstain from or discontinue the use of any laxatives and any prescription and over-the-counter medications or supplements intended to treat constipation from the time of Screening to the end of the study, except as permitted in this protocol.
* Subject must agree to refrain from making any lifestyle changes that may affect IBS-C symptoms from the time of Screening to the end of the study.

Exclusion Criteria:

* Subject has taken IBS treatments (prescription or over-the-counter), proton pump inhibitors, laxatives, antibiotics.
* Subject did not complete Study SB-2-010-001 or more than 7 days have elapsed since the subject's last dose of study drug in that study.
* Subject reports loose (mushy) or watery stools (Bristol Stool Form Scale [BSFS] score of 6 or 7) in the absence of any laxative, or has a BSFS score of 6 for more than 1 spontaneous bowel movement (SBM) or a BSFS score of 7 for any SBM during the last 7 days of diary reporting for Study SB-2-010-001.
* Subject has any abnormal laboratory results, electrocardiogram (ECG) findings, or physical examination findings deemed clinically significant by the investigator at the Study SB-2-010-001 End-of-Study Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Hialeah, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Miami Springs, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Virginia Gardens, Florida
  - West Palm Beach, Florida
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose SYN-010: 21-mg SYN-010
- Placebo: Placebo
Period: Overall Study
Arm/Group | High Dose SYN-010 | Low Dose SYN-010 | Placebo
Started | 17 | 20 | 17
Completed | 16 | 18 | 15
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- 42-mg SYN-010/42-mg SYN-010: 42-mg SYN-010 in study NCT02495623 followed by 42-mg SYN-010 in current study
- 21-mg SYN-010/42-mg SYN-010: 21-mg SYN-010 in study NCT02495623 followed by 42-mg SYN-010 in current study
- Placebo/42-mg SYN-010: Placebo in study NCT02495623 followed by 42-mg SYN-010 in current study
- Total: Total of all reporting groups
Arm/Group | 42-mg SYN-010/42-mg SYN-010 | 21-mg SYN-010/42-mg SYN-010 | Placebo/42-mg SYN-010 | Total
Number analyzed (Participants) | 17 | 20 | 17 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (8.67) | 42.6 (6.30) | 46.4 (11.16) | 44.0 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 13 | 42
  Male | 5 | 3 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Study 1 (NCT02495623) Baseline in the Area Under the Curve (AUC) of Breath CH4 Production, Based on a 180-minute Lactulose Breath Test (LBT) at Day 56 Post-dose.
Time Frame: 56 days
Population: In this table, there are 16, 18 and 14 subjects in the 42mg/42mg, 21mg/42mg and Placebo/42mg group, respectively. This is a change-from-baseline analysis, only subjects with no missing values AT BOTH baseline and Day 56 are included in the analysis, so the number of subjects in each group is less than the number of subjects that started the study.
Measure: Mean (Standard Deviation); unit: ppm*hr
Groups:
- 42-mg SYN-010/42-mg SYN-010: Subjects were on 42 mg in the 4-week (double-blind) study and were continued on 42 mg in the 8-week extension study
- 21-mg SYN-010/42-mg SYN-010: Subjects were on 21 mg in the 4-week (double-blind) study and then received 42 mg in the 8-week extension study
- Placebo/42-mg SYN-010: Subjects were on placebo in the 4-week (double-blind) study and then received 42 mg in the 8-week extension study
Arm/Group | 42-mg SYN-010/42-mg SYN-010 | 21-mg SYN-010/42-mg SYN-010 | Placebo/42-mg SYN-010
Number analyzed (Participants) | 16 | 18 | 14
ppm*hr | 73.78 (70.62) | 63.91 (75.68) | 33.30 (34.23)

ADVERSE EVENTS:
Arm/Group | 42-mg SYN-010/42-mg SYN-010 | 21-mg SYN-010/42-mg SYN-010 | Placebo/42-mg SYN-010
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 2/20 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 42-mg SYN-010/42-mg SYN-010 (N=17) | 21-mg SYN-010/42-mg SYN-010 (N=20) | Placebo/42-mg SYN-010 (N=17)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ALT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood ALP increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood CPK increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood LDH increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators do not see trial results ahead of public disclosure unless it is under CDA. Investigators will not be allowed to publish or disclose any study results prior to sponsor communicating it to the public.